CLINICAL TRIAL: NCT06590259
Title: A Study on the Efficacy and Safety of Multi-mode Ablation Combined With Systemic Therapy Including PD-1 Inhibitor in the Treatment of Colorectal Cancer Liver Metastasis(CRCLM)
Brief Title: A Study on the Efficacy and Safety of Multi-mode Ablation Combined With Systemic Therapy in the Treatment of CRCLM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Zan, Chief of Medical Oncology, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231124
Record Dates: First submitted 2024-05-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer Liver Metastasis
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-mode thermal ablation combined with systemic therapy including PD-1 inhibitor (Experimental): Multi-mode ablation therapy +systemic therapy including PD-1 inhibitor (sintilimab 200 mg IV D1+ mFOLFOX6 or FOLFIRI+bevacizumab or cetuximab（determined according to the subject's first-line chemotherapy regimen), Q3W, chemotherapy for 4-6 cycles. Sintilimab continues until disease progression, not exceeding a maximum of 2 years.)
  Interventions: Device: Multi-mode tumor treatment system; Drug: Sintilimab+mFOLFOX6 or FOLFIRI+bevacizumab or cetuximab

INTERVENTIONS:
Device: Multi-mode tumor treatment system — All subjects are treated using the multi-mode tumor treatment system (Shanghai MAaGI Medical Technology Co., Ltd), with the treatment procedure conducted according to the temperature control mode for tumor ablation. Complete ablation of intrahepatic lesions is achieved to realize an intrahepatic no-evidence-of-disease (NED) state. For lesions that could not be ablated in a single session, two treatments are performed to achieve NED within the liver.
  Other Names: MTT-P1
Drug: Sintilimab+mFOLFOX6 or FOLFIRI+bevacizumab or cetuximab — Systemic therapy including PD-1 inhibitor starts on the 7th day after ablation (sintilimab 200 mg IV D1 + mFOLFOX6 or FOLFIRI + bevacizumab or cetuximab (determined according to the subject's first-line chemotherapy regimen), Q3W, chemotherapy for 4-6 cycles. Sintilimab continues until disease progression, not exceeding a maximum of 2 years.）
  Other Names: Systemic therapy including PD-1 inhibitor

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of multi-mode ablation combined with systemic therapy including PD-1(programmed death receptor 1) inhibitor for colorectal cancer liver metastasis and furthermore to clarify its application value by comparing preoperative and postoperative immune indicators.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective study to evaluate the efficacy and safety of multi-mode ablation combined with systemic therapy including PD-1 inhibitor in the treatment of colorectal cancer liver metastasis. The study includes 20 patients with colorectal cancer liver metastasis that has failed first-line therapy and is unresectable. All patients will receive multi-mode ablation to achieve complete remission of liver lesions followed by systemic therapy including PD-1 inhibitor.

This study will provide preliminary data on the efficacy and safety of multi-mode ablation combined with systemic therapy including PD-1 inhibitor in the treatment of colorectal cancer liver metastasis, which could lead to larger randomized trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, gender not specified;
2. Pathologically or clinically confirmed colorectal cancer liver metastases, with liver lesions unsuitable for surgical resection or intolerance or refusal of surgical resection;
3. In the case of an unresectable primary tumor or recurrence, the absence of serious complications such as bleeding or obstruction;
4. Failure of first-line treatment, with disease progression or new liver metastases;
5. No more than 5 liver lesions, with single lesion diameter ≤ 3cm;
6. For those who have received previous chemotherapy, radiotherapy or local liver treatment, the interval from the last systemic treatment or local liver treatment should be at least 1 month;
7. Child-Pugh A or B; bilirubin ≤ 3.0 mg/dL, creatinine ≤ 2.5 mg/dL, white blood cell count ≥ 2.0 ×10^9/L, platelets ≥ 100 ×10^9/L;
8. ECOG PS ≤ 2;
9. Willing to accept subsequent treatment regimens that include anti-PD-1 monoclonal antibody therapy.

Exclusion Criteria:

1. Liver function Child-Pugh class C;
2. Expected survival < 3 months;
3. Major organ insufficiency or failure;
4. Active infection;
5. Irreversible coagulation disorders;
6. Refractory massive ascites, pleural effusion or cachexia;
7. Unable to cooperate with treatment;
8. Any other factors deemed inappropriate for inclusion or that may affect the subject's participation in the study, as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | max 24 months
  Progression free survival (PFS) is defined as the time from the start of treatment until the criteria for documented progression of disease (or until death due to any cause) are met, whichever comes first according to RECIST 1.1.

SECONDARY OUTCOMES:
Local Progression Free Survival (LPFS) | max 24 months
  Local progression-free survival (LPFS) is defined as the time from the start of treatment until documented local progression of the lesion(s) under assessment, or until death from any cause, whichever comes first according to RECIST 1.1.
Objective Response Rate (ORR) | max 24 months
  Objective response rate (ORR) is defined as the proportion of patients with a complete response or partial response to treatment according to RECIST 1.1.
Overall Survival (OS) | max 24 months
  Overall survival (OS) is defined as the time from the start of treatment until death from any cause.
Rate of adverse events | max 24 months
  The rate of adverse events will be calculated as the number of participants experiencing any adverse event divided by the total number of participants enrolled in the study.
Immune indicator analysis | max 24 months
  Immune indicator analysis will be conducted to evaluate the immune status and response of participants to the intervention. This will include the assessment of various immune cell populations and markers, such as:
  * CD4+ and CD8+ T lymphocyte counts and ratios.
  * Natural Killer (NK) cell activity and counts.
  * B cell counts and subsets.
  * Dendritic cell (DC) counts and functionality.
  * Monocyte counts and subsets.
  * Neutrophil, eosinophil and basophil counts.
  * Myeloid-derived suppressor cell (MDSC) counts. The analysis will utilize flow cytometry to quantify these immune indicators from blood samples collected at specified time points before, during and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chief physician of Medical Oncology, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China